CLINICAL TRIAL: NCT02645825
Title: Analyse du caractère prédictif de l'échographie Ganglionnaire Pour le Diagnostic de bégninité ou malignité d'Une adénopathie Superficielle
Brief Title: Predictive Character Analysis of Ganglionic Echography for the Diagnostic of Benin or Malignant Superficial Adenopathy
Acronym: EGAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EGAS - RB 14.077
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Superficial Adenopathy
Keywords: superficial adenopathy - echography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators need to establish a formal diagnostic of superficial adenopathy through complementary investigations to find etiologic diagnostic ( Echography, adenogram).

Echography examination should be a guide to take in charge the adenopathy and to predict presence of malignant (primitive) or benin (reactional) character of adenopathy. The aim of this study is to codify the management of adenopathic patient with a diagnostic in 48 hours after examination. This fast diagnostic helps to prevent unnecessary biopsy, to avoid wasting time in case of a serious pathology.

ELIGIBILITY:
Inclusion Criteria:

- superficial adenopathy

Exclusion Criteria:

- obvious adenopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from ambulatory medicine consultation with superficial adenopathy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Parameter of echography | inclusion
  The benign or malignant nature of adenopathy (or lymphadenopathy) confirmed by adenogram results +/- lymph node biopsy (as the gold standard)"

CONTACTS AND LOCATIONS:
Overall Officials: Christian Berthou, Principal Investigator — CHRU de Brest
Locations (16):
- France (16):
  - Cabinet Brest, Brest
  - Caninet Brest Centre, Brest
  - CHRU de Brest, Brest
  - Cabinet Ergue Gaberic, Ergue Gaberit
  - Cabinet Ergue Gaberit, Ergue Gaberit
  - Cabinet Ergue Gaberic, Ergué-Gabéric
  - Cabine Le Guivinec, Guilvinec
  - Cabinet Le Guilvinec, Guilvinec
  - Cabinet Lamneur, Lanmeur
  - Cabinet Lanmeur, Lanmeur
  - Cabinet Brest Centre, Le Relecq-Kerhuon
  - Cabinet Lesconil, Lesconil
  - Cabinet Penmarch, Penmarch
  - Cabinet Plouegat Guerrand, Plouegat Guerrand
  - Cabinet Quimper, Quimper
  - CHIC Quimper, Quimper